CLINICAL TRIAL: NCT03934762
Title: Effect of Aloe Vera Ointment Application on Muscle Damage and Performance Recovery Kinetics Following an Intense Eccentric Exercise Protocol: A Pilot Study.
Brief Title: Aloe Vera Ointment Application and Skeletal Muscle Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ALOE VERA-PILOT STUDY-UTH
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-04

CONDITIONS: Skeletal Muscle Damage; Exercise-induced Aseptic Inflammation; Performance
Keywords: aseptic inflammation; muscle trauma; muscle strength; aloe vera

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Active Comparator): A placebo solution will be applied on the quadriceps of one of the lower limbs immediately after the exercise protocol and daily for 7 consecutive days.
  Interventions: Biological: Placebo
- Natural aloe vera (Experimental): A natural aloe vera solution (peel and leaf) will be applied on the quadriceps of one of the lower limbs immediately after the exercise protocol and daily for 7 consecutive days.
  Interventions: Biological: Natural Aloe Vera
- Aloe vera soup (Experimental): An aloe vera soup solution will be applied on the quadriceps of one of the lower limbs immediately after the exercise protocol and daily for 7 consecutive days.
  Interventions: Biological: Aloe vera soup

INTERVENTIONS:
Biological: Placebo — A placebo solution that will not include aloe vera will be applied on the quadriceps of one of the lower limbs.
  Arms: Placebo
Biological: Natural Aloe Vera — Natural aloe vera solution including peel and leaf from aloe will be applied on the the quadriceps of one of the lower limbs.
  Arms: Natural aloe vera
Biological: Aloe vera soup — Aloe vera solution including aloe vera soup will be applied on the the quadriceps of one of the lower limbs.
  Arms: Aloe vera soup

SUMMARY:
Aloe vera, sometimes described as pharmaceutical aloe, is a flowering succulent plant with many therapeutic properties such as wound and burn wound healing, treatment of diabetes and reduction of blood lipid profile. These benefits have been primary attributed to its high content in polysaccharides, anthraquinones and lectins. However, aloe vera includes more than 200 ingredients and nutrients (i.e. vitamins, saponins, amino acids, anthraquinones, minerals and trace-elements, salicylic acid, saccharides, lignin, enzymes, sterols) the combination of which offers more powerful effects and health-related benefits compared to each one of them separately. Thus, based on the ingredients and nutrients included, it has been proposed that aloe vera may also offer anti-inflammatory, antioxidative, analgesic and anabolic benefits.

Exercise training, especially when it is unaccustomed or characterized by increased intensity, results in skeletal muscle microtrauma accompanied by elevated plasma levels of Creatine Kinase (CK), increased sensation of muscle soreness (DOMS), reduced force generating capacity and marked declines in speed and agility. Both anti-inflammatory and antioxidative mechanisms in skeletal muscle are crucial for the termination of inflammatory response and muscle healing process following exercise-induced aseptic muscle injury and inflammation.

Although, it has been proposed that ale vera may elicit anti-inflammatory and antioxidative activity, its effectiveness in alleviating exercise-induced skeletal muscle injury and its symptoms, has not been investigated yet. Therefore, the aim of the present pilot study is to examine the effect of transdermal aloe veral delivery on skeletal muscle damage symptoms following an intense eccentric exercise protocol.

DETAILED DESCRIPTION:
For the purpose of study, ten male participants will be included in a pilot clinical trial.

Initially, participants will undergo a baseline testing including assessment of body height, body mass and body composition, isokinetic evaluation of isometric, concentric and eccentric muscle strength of quadriceps, determination of VO2max, evaluation of DOMS level and resting blood sampling for the measurement of CK. Participants will be also provided with 7-day diet recalls and will be taught by a trained dietitian on how to adjust food/liquid portions and sizes and how to complete diet recalls (1 recall/day over a 7-day period).

After baseline testing, subjects will participate in two trials, in a randomized, double-blind repeated measures design. In the first trial they will execute a bilateral eccentric exercise protocol. Immediately after the exercise protocol and daily for 7 consecutive days, will be applied transdermal treatment with placebo (Control) in one leg and with natural aloe vera (Experimental, aloe vera peel and leaf) in the other. Following a 7-day wash-out period the second trial will be conducted. Participants will execute the same eccentric exercise protocol, but they will be treated with either placebo (Control) or aloe vera soup (Experimental). The selection of the treatment for each leg will be randomly selected. In both trials, assessment of DOMS and strength (isometric, concentric and eccentric) in both legs and blood sampling (for the measurement of CK) will be performed at 1h and 6h post-exercise as well as daily for 7 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Absence of musculoskeletal injury for at least 6 months prior to the study.
* No consumption of performance-enhancing supplements or medication for at least 6 months prior to the study.
* No consumption of anti-inflammatory and antioxidant supplements for at least 6 months prior to the study.
* No participation in exercise including eccentric muscle contractions for at least 3 days prior to the study.

Exclusion Criteria:

* Recent history of musculoskeletal injury.
* Consumption of performance-enhancing supplements and medication.
* Consumption of anti-inflammatory and antioxidant supplements (> 6 months).
* Participation in exercise including eccentric muscle contractions during the last 3 days prior to the study.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change in creatine kinase activity in plasma | At baseline, 1 hour post-exercise, 6 hours post-exercise and daily for 7 consecutive days post-exercise
  Creatine kinase activity will be measured in plasma by utilizing a Clinical Chemistry Analyzer and commercially available kits.
Change in performance of knee extensor muscles | At baseline, 1 hour post-exercise, 6 hours post-exercise and daily for 7 consecutive days post-exercise
  Maximal knee extensor concentric, eccentric and isometric peak torque will be measured on an isokinetic dynamometer.
Change in delayed onset of muscle soreness | At baseline, 1 hour post-exercise, 6 hours post-exercise and daily for 7 consecutive days post-exercise
  Muscle soreness will be assessed during palpation of the muscle belly and the distal region of relaxed quadriceps muscle following three repetitions of a full squat.

CONTACTS AND LOCATIONS:
Locations (1):
- SmArT LABORATORY, SCHOOL OF PHYSICAL EDUCATION & SPORTS SCIENCES, UNIVERSITY OF THESSALY, Trikala, Greece